CLINICAL TRIAL: NCT05380895
Title: Comparison of Daytime Surgery in Varicose Veins Patients With and Without Superficial Venous Thrombosis: a Propensity Score Matched Analysis
Brief Title: Comparison of Daytime Surgery in Varicose Veins Patients With and Without Superficial Venous Thrombosis
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Sun Yat-Sen Memorial Hospital of Sun Yat-Sen University (Other)
Responsible Party: Sponsor
Other Study IDs: SYSKY-2022-013-01
Record Dates: First submitted 2022-05-08; First posted 2022-05-19 (Actual); Last update posted 2022-05-19 (Actual); Status verified 2022-05

CONDITIONS: Varicose Veins; Superficial Venous Thrombosis; Day Surgery
MeSH Terms: conditions — Varicose Veins

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- SVT group: Varicose vein patients complicated with superficial thrombophlebitis
- Non-SVT group: Patients had varicose vein only

SUMMARY:
Varicose veins of lower extremities are the most common disease in vascular surgery, and daytime surgery has gradually become the mainstream of varicose veins of lower extremities. Superficial venous thrombosis is one of the common complications of varicose veins of lower limbs. Current consensus is that patients with superficial venous thrombosis should be treated with standardized anticoagulant therapy to prevent their progression to venous thrombotic disease.SVT patients need standardized anticoagulant therapy for a period of time, while DS is current mainstream treatment of VV. Will the existence of SVT affect the safety and efficacy of DS of VV, leading a need of changing the treatment strategy and carrying out anticoagulant treatment for SVT before DS on VV patients? To date, there is no research on this issue. Therefore, we conducted this study to comprehensively evaluate the safety, feasibility, perioperative and long-term efficacy of DS in VV patients complicated with SVT, and systematically compared patients who had VV only.

DETAILED DESCRIPTION:
Varicose veins （VV） of lower extremities are common diseases in outpatient and inpatients. Approximately 25% of the world's adult population suffer from varicose veins of lower extremities, of which, the prevalence of VV in China reaches 8.9%, affecting more than 100 million people. From this, VV is a highly prevalent disease and one of the major public health problems in the world, placing huge economic and medical burden on both patients and health care.

Unlike inpatient surgery (IS), by which previous VV patients were mainly treated, Day surgery (DS), also known as ambulatory surgery，tends to exhibit higher medical efficacy and less cost of health care. Moreover, the development of endovenous treatment and sclerotherapy technology makes it feasible for clinicians to treat VV through DS. DS for VV patients can well alleviate the contradiction between the growth of medical demand and the shortage of medical resources, considering the fact that merely 4.3 beds are available per 1000 people on average in China.

Superficial venous thrombosis (SVT) of lower extremities, as a common complication of VV, is characterized by pain, erythema and usually palpable nodular mass of the diseased veins. Currently, VV still are the most common risk factor of SVT, despite SVT can exist independently. Previous studies have shown that the probability of SVT in VV patients ranges from 4% to 59%, while up to 80% of SVT patients are complicated with VV. SVT used to be considered as a self-limiting benign disease lacking in enough attention in clinical decision-making. However current researches show that SVT is closely related to the occurrence of venous thromboembolism (VTE), and especially when SVT involves the blood vessels connecting the deep venous system, the probability of VTE is as high as 18%, which seriously threatens the safety of patients. Due to the close relationship between SVT and VTE, the treatment of SVT is gaining its importance recent years. The latest guidelines of CHEST recommend 45 days of anticoagulant therapy for patients with SVT to reduce their risk of progressing to VTE, and surgery, including ligation of the great saphenofemoral joint or stripping of the superficial vein of thrombosis, is also applied in the treatment of SVT. SVT patients need standardized anticoagulant therapy for a period of time, while DS is current mainstream treatment of VV. Will the existence of SVT affect the safety and efficacy of DS of VV, leading a need of changing the treatment strategy and carrying out anticoagulant treatment for SVT before DS on VV patients? To date, there is no research on this issue.

It remains unclear whether the combination of SVT will have a negative impact on the DS of VV patients. Therefore, we conducted this study to comprehensively evaluate the safety, feasibility, perioperative and long-term efficacy of DS in VV patients complicated with SVT, and systematically compared patients who had VV only. To reduce the possible selection bias, a propensity score matching model (PSM) was used to balance the baseline data of the two groups of patients.

ELIGIBILITY:
Inclusion Criteria:

* VV patients with the CEAP grade of C2-C5;
* At the age 18 to 75;
* Treated by day surgery

Exclusion Criteria:

* Patient has a history of DVT or is suffering from DVT;
* Patients with liver and renal failure;
* Patients in hypercoagulable state；
* Patients with anticoagulant therapy before operation;
* Patients with active ulcer；
* Patient is intolerant to foam sclerotherapy

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This is a single center retrospective cohort study, which retrospectively analyzed the clinical data of VV patients treated in Sun Yat-sen Memorial Hospital of Sun Yat-sen University from 2015 to 2021. Doppler ultrasound, combined with clinical examination, was used in the diagnosis of SVT.
Sampling Method: Non-Probability Sample
Enrollment: 699 (Estimated)
Dates: Start 2022-06-10 (Estimated); Primary Completion 2024-06-10 (Estimated); Study Completion 2025-06-10 (Estimated)

PRIMARY OUTCOMES:
postoperative deep venous thrombosis | Events within one week after surgery
  deep venous thrombosis after surgery
saphenous nerve injury | Events during surgery
  saphenous nerve injury after surgery
subcutaneous induration | Events within one week after surgery
  subcutaneous induration after surgery

SECONDARY OUTCOMES:
varicose veins recurrence | recurrence within 12 months follow-up after surgery
  VV recurred during follow-up
superficial venous thrombosis formation | Events within 12 months follow-up after surgery
  superficial venous thrombosis formatted during follow-up
deep venous thrombosis | Events within 12 months follow-up after surgery
  deep venous thrombosis event during follow-up
skin burns | Events during surgery
  skin burns after operation
bleeding requiring intervention | Events during surgery
  bleeding requiring intervention during operation

CONTACTS AND LOCATIONS:
Overall Officials: Huang Kai, doctor, Study Chair — Sun Yat-Sen Memorial Hospital of Sun Yat-Sen University
Locations (1):
- Sun Yat-sen Memorial Hospital, Sun Yat-sen University, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No
Clinical treatment information that does not design patient privacy

REFERENCES:
- [Derived] Xu J, Xu X, Tian J, Huang M, Xia Z, Luo X, Zheng J, Huang K. Comparison of day surgery between varicose veins with and without superficial venous thrombosis below knee: a propensity score-matched analysis. BMC Cardiovasc Disord. 2023 Aug 3;23(1):387. doi: 10.1186/s12872-023-03398-2. PMID 37537563